CLINICAL TRIAL: NCT01357694
Title: Open Monocentric Randomized Clinical Trial on the Efficacy of the Psychotherapeutic Bridging Intervention in Anesthesiology (BRIA)
Brief Title: BRIA - Bridging Intervention in Anesthesiology
Acronym: BRIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRIA
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Psychiatric or Mood Diseases or Conditions
Keywords: psychotherapy; depression; anxiety; surgical patients
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- psychotherapeutic contacts (Experimental)
  Interventions: Behavioral: psychotherapeutic contacts
- control group (No Intervention)

INTERVENTIONS:
Behavioral: psychotherapeutic contacts — psychotherapeutic contacts during inpatient hospital stay and up to 3 months outpatient appointments after discharge
  Arms: psychotherapeutic contacts

SUMMARY:
The major purpose of this study is to determine whether psychotherapeutic contacts for surgical patients with psychological distress are an effective treatment during the postoperative period to improve the rate of treatment participation in subsequent psychosocial treatment programs.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the efficacy of psychotherapeutic contacts that aim at motivating and supporting surgical patients with psychiatric disorders in participating in subsequent psychosocial treatment options like psycho- and addiction therapy (RCT). The secondary objective is to investigate whether preoperatively assessed psychosocial factors are associated with surgical outcomes (preoperative computer-assisted self assessment).

The Bridging Intervention in Anesthesiology (BRIA) has been designed as a feasible treatment option to reach patients from all surgical fields. Implemented in the preoperative anesthesiological assessment clinic this therapy program comprises two major elements: (1) A computer assisted self assessment of social, lifestyle and psychological factors including a comprehensive battery of psychiatric screening tests; (2) Psychotherapeutic contacts with the objective to motivate patients with psychiatric disorders and support them in participating in subsequent psychosocial treatment programs. The self assessment will be offered to all adult surgical patients of the preoperative anesthesiological assessment clinic during inclusion period (current 5104 patients). Data on surgical outcomes will be collected prospectively during a 6-month-follow-up, and regression analyses will be performed to determine the extent of associations between psychosocial factors and outcomes. Patients with clinically relevant psychological distress (i.e. scoring above the cut-off of one of applied standardized screening questionnaires) will be offered to participate in the RCT on the psychotherapy part of BRIA (220 patients). Data on primary and secondary outcomes will be collected 6 months and 24 months, respectively, after baseline assessment.

ELIGIBILITY:
Inclusion and exclusion criteria for participating at the preoperative computer-assisted self assessment were defined as follows:

Inclusion criteria:

* Written informed consent to participate in the first part of study after having been properly instructed
* patient of the preoperative anesthesiological assessment clinic
* age ≥18 years.

Exclusion criteria:

* Surgery with an emergency or urgent indication
* inability to attend the preoperative assessment clinic (bedside visit)
* insufficient knowledge of German language
* members of the hospital staff
* admitted in police custody
* accommodation in an institution by official or court order
* being under guardianship
* psychiatric, neurological or other condition associated with limited legal capability or limited capability of being properly instructed or giving informed consent.

Additional inclusion and exclusion criteria of the RCT (Enrollment: 220 patients) were defined as follows:

Inclusion criteria:

* Written informed consent to participate in the RCT after having been properly instructed
* acute significant psychiatric distress (scoring above of at least one of the cut-off values of WHO-5, PHQ-2, GAD-2, HADS-D, HADS-A, AUDIT) and/or being tobacco smoker, and/or having consumed illicit drugs during the last 12 months.

Exclusion criteria:

* Acute severe psychiatric condition (acute episode of psychotic disorder, severe substance use disorder including serious withdrawal symptoms)
* severe acute suicidality
* homelessness
* participation in a psychopharmacological clinical trial at baseline assessment or 1 month before, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
participation in psychosocial therapy | six months after baseline assessment
  rate of patients who participate in succeeding outpatient or inpatient psychosocial treatment (psychotherapy, addiction therapy)

SECONDARY OUTCOMES:
psychiatric distress | 6 months after baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Claudia D Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine, Charité - Universitätsmedizin Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Charité - Universitätsmedizin Berlin, Germany, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Krampe H, Goerling U, Spies CD, Gerhards SK, Enge S, Salz AL, Kerper LF, Schnell T. Sense of coherence, mental well-being and perceived preoperative hospital and surgery related stress in surgical patients with malignant, benign, and no neoplasms. BMC Psychiatry. 2020 Nov 27;20(1):567. doi: 10.1186/s12888-020-02953-x. PMID 33246438
- [Derived] Krampe H, Barth-Zoubairi A, Schnell T, Salz AL, Kerper LF, Spies CD. Social Relationship Factors, Preoperative Depression, and Hospital Length of Stay in Surgical Patients. Int J Behav Med. 2018 Dec;25(6):658-668. doi: 10.1007/s12529-018-9738-8. PMID 30105602
- [Derived] Krampe H, Salz AL, Kerper LF, Krannich A, Schnell T, Wernecke KD, Spies CD. Readiness to change and therapy outcomes of an innovative psychotherapy program for surgical patients: results from a randomized controlled trial. BMC Psychiatry. 2017 Dec 29;17(1):417. doi: 10.1186/s12888-017-1579-5. PMID 29284443